CLINICAL TRIAL: NCT05844995
Title: An Open-label, Single-dose, Pharmacokinetic Study of Acetaminophen/Naproxen Sodium Fixed Combination Tablets in Adolescents 12 to <17 Years of Age With Orthodontic Pain
Brief Title: A Study of Acetaminophen/Naproxen Sodium Fixed Combination Tablets in Adolescents 12 to <17 Years of Age With Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCSPAP005203; CCSPAP005203 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Orthodontic Pain
MeSH Terms: interventions — Acetaminophen; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acetaminophen /Naproxen Sodium (Experimental): Participants with age group 12 to less than (<) 17 years who undergone a non-surgical orthodontic procedure will enroll and receive fixed dose combination of acetaminophen/naproxen sodium tablet orally on baseline (Day 0).
  Interventions: Drug: Acetaminophen/Naproxen Sodium

INTERVENTIONS:
Drug: Acetaminophen/Naproxen Sodium — Fixed dose combination of acetaminophen/naproxen sodium tablet will be administered orally.

SUMMARY:
The purpose of this study is to investigate the population pharmacokinetics of acetaminophen and naproxen from a novel acetaminophen /naproxen sodium fixed combination tablet in adolescents 12 to less than (<) 17 years of age with post-procedure orthodontic pain and to describe the effect of subject-specific covariates, including age and body weight, on inter-subject variability in acetaminophen and naproxen pharmacokinetics in adolescents 12 to <17 years of age with post-procedure orthodontic pain.

ELIGIBILITY:
Inclusion Criteria:

* A parent or a legal guardian of the participant has signed and dated the informed consent document and a written assent has been signed by the participant
* Has undergone an orthodontic procedure within 72 hours prior to dosing
* Is otherwise a healthy adolescent between the ages of 12 to less than (<) 17 years at baseline (dosing). Health is defined as the absence of clinically relevant abnormalities as judged by the principle investigator (PI) on the basis of a detailed medical history, physical examination, blood pressure, respiratory rate and pulse rate measurements, and clinical laboratory tests. The responsible PI may request additional investigations or analyses if necessary
* Has a minimum weight of 72 pounds and has a Body Mass Index (BMI) between the 5th and 95th percentile for their age at dosing
* Has been fasted for at least 10 hours prior to dose administration of the investigational product
* Is a non-tobacco user or previous user who completely stopped smoking or using any form of tobacco or nicotine-containing product [including e-cigarettes, cigarettes, non-combusted cigarettes, cigars, smokeless tobacco (such as dip, snuff, snus, and chewing tobacco)] for at least 12 months before screening visit of this study
* If female, have a negative test for pregnancy at screening and baseline (dosing)
* Females of childbearing potential and males agree to the contraceptive requirements
* Is able to comprehend the requirements of the study (based upon clinical site personnel's assessment) and is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified within the protocol
* Are willing for investigational product of this study to be the only analgesic product used during the study

Exclusion Criteria:

* Use of prescription or non-prescription medications within a period less than 5 half-lives before the first investigational product (IP) administration unless these are contraceptives or occasional use of other medications approved by the Investigator
* Use of Ibuprofen within 6 hours prior to the dose administration of the investigational product
* Use of any vitamins, dietary and herbal supplements within seven days before first dose of study drug
* Has hypersensitivity to acetaminophen, naproxen, other non-steroidal anti-inflammatory drug (NSAIDs), including acetylsalicylic acid, or to any of the ingredients
* If female, has a positive pregnancy test or is breast-feeding or currently trying to become pregnant
* Has a positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV)
* Has a positive test for drugs of abuse at screening or baseline (dosing)
* Has difficult venipuncture access and/or refuses to undergo venipuncture
* Has clinically significant renal or hepatic impairment according to the medically qualified Investigator discretion, or presence of a disease, which in the opinion of the Investigator, would preclude the use of IP
* Has a history of peptic ulcers, gastrointestinal bleeding of any etiology, bleeding disorders, gastrointestinal disease (including chronic heartburn or gastroesophageal reflux disease, or any other active inflammatory disease of the gastrointestinal tract such as ulcerative colitis or crohn's disease), or has a history of gastrointestinal surgery (including cholecystectomy) that would affect the pharmacokinetic (PK) assessment of the drug or the safety of the participant
* Has history of substance abuse, as judged by the PI, within 12 months preceding this study
* Has used alcohol within 24 hours of baseline visit and/or has positive alcohol test in expired air at screening or baseline visit
* Has used food or beverages containing xanthines (that is, tea, coffee, cola drinks, energy drinks or chocolate) for 48 hours prior to the dosing and during the study period
* Has used grapefruit and savoy oranges for 48 hours prior to the dosing and during the study period
* Participating in a clinical trial and/or treated with any investigational product within 3 months preceding the dose of study drug
* Has preplanned surgery, procedures, or personal commitments that would interfere with the conduct of the study
* Had an acute blood loss of 50 milliliter (mL) to 249 mL within the 30 days, or 250 mL to 449 mL within the 45 days, or greater than or equal to (>=) 450 mL within the 60 days before first dose administration
* Has any acute or chronic medical or psychiatric condition(s) that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the medically qualified Investigator, would make the participant inappropriate for entry into this study
* Has any clinically important abnormal value for serum chemistry, hematology, or urinalysis at screening. Laboratory values will generally be within the normal ranges, although minor deviations in tests (except those explicitly specified in the inclusion criteria) that are not considered clinically important by the Investigator are acceptable
* Is related to persons involved directly or indirectly with the conduct of the study (that is, principal investigator, sub-investigators, study coordinators, other study personnel, employees or contractors of the Sponsor or Johnson & Johnson (J&J) subsidiaries, and the family of each)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Apparent Clearance (CL/F) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  CL/F is defined as apparent clearance of acetaminophen/naproxen sodium.
Apparent Central Volume of Distribution (Vc/F) After Oral Dosing of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Vc/F is defined as apparent central volume of distribution after oral dosing of acetaminophen/naproxen sodium.
Apparent Peripheral Volume of Distribution (Vp/F) After Oral Dosing of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Vp/F is defined as apparent peripheral volume of distribution after oral dosing of acetaminophen/naproxen sodium.
Apparent Inter-compartmental Clearance (Q/F) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Q/F is defined as apparent inter-compartmental clearance of acetaminophen/naproxen sodium.
First-order Absorption Rate Constant (Ka) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Ka is defined as first-order absorption rate constant of acetaminophen/naproxen sodium.
Maximum Plasma Concentration (Cmax) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Cmax is defined as maximum plasma concentration of acetaminophen/naproxen sodium.
Time of occurrence of Maximum Plasma Concentration (Tmax) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Tmax is defined as time of occurrence of maximum plasma concentration of acetaminophen/naproxen sodium.
Area Under the Plasma Concentration versus Time Curve from Start of Drug Administration Until the Time of the Last Measurable Plasma Concentration (AUC[0-t]) | Pre-dose up to 48 hours post dose
  AUC(0-t) is defined as area under the plasma concentration versus time curve from start of drug administration until the time of the last measurable plasma concentration of acetaminophen/naproxen sodium.
Area Under the Plasma Concentration versus Time Curve From Start of Drug Administration Until Infinity (AUC[0-infinite]) | Pre-dose up to 48 hours post dose
  AUC(0-infinite) is defined as area under the plasma concentration versus time curve from start of drug administration until infinity of acetaminophen/naproxen sodium.
Terminal Elimination Rate Constant (lambda[z]) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  Lambda(z) is defined as terminal elimination rate constant of acetaminophen/naproxen sodium.
Half Life (t1/2) of Acetaminophen/Naproxen Sodium | Pre-dose up to 48 hours post dose
  T1/2 is defined as half life of acetaminophen/naproxen sodium.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 3 days
  An AE is any untoward medical occurrence that occurs in participants after they have signed an informed consent for the study. The event does not need to have a suspected causal relationship with the investigational product (IP).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Consumer Inc. (J&JCI) Clinical Trial, Study Director — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- JBR Clinical Research LLP, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] GUZMAN F, BRAUN C, LIM RK, POTTER GD, RODGERS DW. NARCOTIC AND NON-NARCOTIC ANALGESICS WHICH BLOCK VISCERAL PAIN EVOKED BY INTRA-ARTERIAL INJECTION OF BRADYKININ AND OTHER ALGESIC AGENTS. Arch Int Pharmacodyn Ther. 1964 Jun 1;149:571-88. No abstract available. PMID 14191090
- [Background] LIM RK, GUZMAN F, RODGERS DW, GOTO K, BRAUN C, DICKERSON GD, ENGLE RJ. SITE OF ACTION OF NARCOTIC AND NON-NARCOTIC ANALGESICS DETERMINED BY BLOCKING BRADYKININ-EVOKED VISCERAL PAIN. Arch Int Pharmacodyn Ther. 1964 Nov 1;152:25-58. No abstract available. PMID 14248351
- [Background] Aronoff DM, Oates JA, Boutaud O. New insights into the mechanism of action of acetaminophen: Its clinical pharmacologic characteristics reflect its inhibition of the two prostaglandin H2 synthases. Clin Pharmacol Ther. 2006 Jan;79(1):9-19. doi: 10.1016/j.clpt.2005.09.009. No abstract available. PMID 16413237
- [Background] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905
- [Background] Mallet C, Daulhac L, Bonnefont J, Ledent C, Etienne M, Chapuy E, Libert F, Eschalier A. Endocannabinoid and serotonergic systems are needed for acetaminophen-induced analgesia. Pain. 2008 Sep 30;139(1):190-200. doi: 10.1016/j.pain.2008.03.030. Epub 2008 May 15. PMID 18485596
- [Background] McGilveray IJ, Mattok GL, Fooks JR, et al. Acetaminophen II: A comparison of the physiological availabilities of different commercial dosage forms. Can J Pharmaceut Sci 1971;6:38-42.
- [Background] Liu DJ, Collaku A, Youngberg SP. Bioavailability and pharmacokinetic profile of a newly-developed twice-a-day sustained-release paracetamol formulation. Int J Clin Pharmacol Ther. 2015 Feb;53(2):172-81. doi: 10.5414/CP202146. PMID 25500485
- [Background] Paracetamol. In: Sweetman S, ed. Martindale - The Complete Drug Reference. London, UK: The Pharmaceutical Press. 37th ed. 2011:76-79.
- [Background] Grosser T, Smyth E, FitzGerald. Anti-Inflammatory, Antipyretic, and Analgesic Agents; Pharmacotherapy of Gout. In: Goodman LS, Brunton LL, Chabner B, Knollman BC. Goodman and Gilman's The Pharmacological Basis of Therapeutics. 12th ed. New York, McGraw-Hill. 2011:959- 1004.
- [Background] McNeil Consumer & Specialty Pharmaceuticals Clinical Pharmacology Report for Protocol 02- 161: Tolerability and multiple-dose pharmacokinetics of acetaminophen (paracetamol) at and above the currently recommended dose. Fort Washington, PA. McNeil Consumer & Specialty Pharmaceuticals Company. Aug 2005.
- [Background] McNeil Consumer Products Company Statistical Report 7: Interim statistical analysis of the study of the bioavailability and antipyretic effectiveness of acetaminophen in children. Fort Washington, PA. McNeil Consumer Products Company. Dec 1978. [Meta-Analysis Code P00102]
- [Background] McNeil Consumer Products Company Statistical Report 65 for Protocol 0-220: A double-blind multiple-dose study of the comparative antipyretic effectiveness and safety of standard and double standard doses of acetaminophen in febrile children. Fort Washington, PA. McNeil Consumer Products Company. Jun 1986. [Meta-Analysis Code P80220]
- [Background] McNeil Protocol 2-227 Data Listings. A double-blind study of the comparative antipyretic effectiveness and safety of a single 15 mg/kg, 30 mg/kg or 40 mg/kg dose of acetaminophen. Oct 1982 [Meta-Analysis Code P82227]
- [Background] McNeil Consumer Products Company Report for Protocol 93-308: Pharmacokinetic and pharmacodynamic modeling of acetaminophen in febrile children: Evaluation of three products. Fort Washington, PA. McNeil Consumer Products Company. 1994. [Meta-Analysis Code P93308]
- [Background] McNeil Consumer Products Company Data Listings for Protocol 1-224: A double-blind study of the comparative antipyretic effectiveness and safety of a single 10 mg/kg, 20 mg/kg or 30 mg/kg dose of acetaminophen. Sep 1981. [Meta-Analysis Code P81224]
- [Background] Ji P, Wang Y, Li Z, Doddapaneni S, Hertz S, Furness S, Sahajwalla CG. Regulatory review of acetaminophen clinical pharmacology in young pediatric patients. J Pharm Sci. 2012 Dec;101(12):4383-9. doi: 10.1002/jps.23331. Epub 2012 Oct 16. PMID 23073837
- [Background] Wilson JT, Brown RD, Bocchini JA Jr, Kearns GL. Efficacy, disposition and pharmacodynamics of aspirin, acetaminophen and choline salicylate in young febrile children. Ther Drug Monit. 1982;4(2):147-80. doi: 10.1097/00007691-198206000-00003. No abstract available. PMID 6980501
- [Background] Levy G. Comparative pharmacokinetics of aspirin and acetaminophen. Arch Intern Med. 1981 Feb 23;141(3 Spec No):279-81. doi: 10.1001/archinte.141.3.279. PMID 7469620
- [Background] Milligan TP, Morris HC, Hammond PM, Price CP. Studies on paracetamol binding to serum proteins. Ann Clin Biochem. 1994 Sep;31 ( Pt 5):492-6. doi: 10.1177/000456329403100512. PMID 7832576
- [Background] Forrest JA, Clements JA, Prescott LF. Clinical pharmacokinetics of paracetamol. Clin Pharmacokinet. 1982 Mar-Apr;7(2):93-107. doi: 10.2165/00003088-198207020-00001. PMID 7039926
- [Background] Paracetamol In: Dollery C., editor. Therapeutic drugs. 2nd ed. Vol 2. Edinburgh: Churchill Livingstone. 1999
- [Background] Peterson RG, Rumack BH. Pharmacokinetics of acetaminophen in children. Pediatrics. 1978 Nov;62(5 Pt 2 Suppl):877-9. PMID 364399
- [Background] Davies NM, Anderson KE. Clinical pharmacokinetics of naproxen. Clin Pharmacokinet. 1997 Apr;32(4):268-93. doi: 10.2165/00003088-199732040-00002. PMID 9113437
- [Background] Product Monograph for Aleve (Naproxen Sodium Tablets USP/Liquid Gels/Capsules 220 mg). Bayer Inc. Consumer Care. Revised January 8th, 2015.
- [Background] Todd PA, Clissold SP. Naproxen. A reappraisal of its pharmacology, and therapeutic use in rheumatic diseases and pain states. Drugs. 1990 Jul;40(1):91-137. doi: 10.2165/00003495-199040010-00006. PMID 2202585
- [Background] Segre EJ. Naproxen sodium (Anaprox): pharmacology, pharmacokinetics and drug interactions. J Reprod Med. 1980 Oct;25(4 Suppl):222-5. PMID 7001021
- [Background] Sevelius H, Runkel R, Segre E, Bloomfield SS. Bioavailability of naproxen sodium and its relationship to clinical analgesic effects. Br J Clin Pharmacol. 1980 Sep;10(3):259-63. doi: 10.1111/j.1365-2125.1980.tb01753.x. PMID 7437243
- [Background] Setiawati S et al. Bioequivalence study with two naproxen sodium tablet formulations in healthy subjects. J Bioequival Availab 2009;1: 28-33.
- [Background] Inc., P., PRODUCT MONOGRAPH, PEDIAPHARM NAPROXEN SUSPENSION, naproxen, 25 mg/mL Suspension, USP, Non-Steroidal Anti-Inflammatory Drug (NSAID) 2018.
- [Background] Valitalo P, Kumpulainen E, Manner M, Kokki M, Lehtonen M, Hooker AC, Ranta VP, Kokki H. Plasma and cerebrospinal fluid pharmacokinetics of naproxen in children. J Clin Pharmacol. 2012 Oct;52(10):1516-26. doi: 10.1177/0091270011418658. Epub 2011 Nov 8. PMID 22067196
- [Background] Altman RD. A rationale for combining acetaminophen and NSAIDs for mild-to-moderate pain. Clin Exp Rheumatol. 2004 Jan-Feb;22(1):110-7. PMID 15005014
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Mehlisch DR, Aspley S, Daniels SE, Southerden KA, Christensen KS. A single-tablet fixed-dose combination of racemic ibuprofen/paracetamol in the management of moderate to severe postoperative dental pain in adult and adolescent patients: a multicenter, two-stage, randomized, double-blind, parallel-group, placebo-controlled, factorial study. Clin Ther. 2010 Jun;32(6):1033-49. doi: 10.1016/j.clinthera.2010.06.002. PMID 20637958
- [Background] Palma-Aguirre JA, Villalpando-Hernandez J, Novoa-Heckel G, Oliva I, Carino L, Lopez-Bojorquez E, Burke-Fraga V, Namur S, Gonzalez-de la Parra M. Bioavailability of two oral-tablet and two oral-suspension formulations of naproxen sodium/paracetamol (acetaminophen): single-dose, randomized, open-label, two-period crossover comparisons in healthy Mexican adult subjects. Clin Ther. 2009 Feb;31(2):399-410. doi: 10.1016/j.clinthera.2009.02.002. PMID 19302912
- [Background] Topolski F, Moro A, Correr GM, Schimim SC. Optimal management of orthodontic pain. J Pain Res. 2018 Mar 16;11:589-598. doi: 10.2147/JPR.S127945. eCollection 2018. PMID 29588616
- [Background] Cheng C, Xie T, Wang J. The efficacy of analgesics in controlling orthodontic pain: a systematic review and meta-analysis. BMC Oral Health. 2020 Sep 18;20(1):259. doi: 10.1186/s12903-020-01245-w. PMID 32948150
- [Background] Monk AB, Harrison JE, Worthington HV, Teague A. Pharmacological interventions for pain relief during orthodontic treatment. Cochrane Database Syst Rev. 2017 Nov 28;11(11):CD003976. doi: 10.1002/14651858.CD003976.pub2. PMID 29182798
- [Background] Krishnan V. Orthodontic pain: from causes to management--a review. Eur J Orthod. 2007 Apr;29(2):170-9. doi: 10.1093/ejo/cjl081. PMID 17488999
- [Background] Polat O, Karaman AI, Durmus E. Effects of preoperative ibuprofen and naproxen sodium on orthodontic pain. Angle Orthod. 2005 Sep;75(5):791-6. doi: 10.1043/0003-3219(2005)75[791:EOPIAN]2.0.CO;2. PMID 16279825
- [Background] Zarif Najafi H, Oshagh M, Salehi P, Babanouri N, Torkan S. Comparison of the effects of preemptive acetaminophen, ibuprofen, and meloxicam on pain after separator placement: a randomized clinical trial. Prog Orthod. 2015;16:34. doi: 10.1186/s40510-015-0104-y. Epub 2015 Oct 14. PMID 26467790
- [Background] Gritsiuk AI. [On the problem of the effect of prednisolone and salicylates on the fibrinolytic activity of the blood in patients with rheumatism]. Ter Arkh. 1967 Sep;39(9):60-1. No abstract available. Russian. PMID 5611706
- [Background] Harrington JT, Isner JM, Kassirer JP. Our national obsession with potassium. Am J Med. 1982 Aug;73(2):155-9. doi: 10.1016/0002-9343(82)90171-1. No abstract available. PMID 7051823
- [Background] Bernhardt MK, Southard KA, Batterson KD, Logan HL, Baker KA, Jakobsen JR. The effect of preemptive and/or postoperative ibuprofen therapy for orthodontic pain. Am J Orthod Dentofacial Orthop. 2001 Jul;120(1):20-7. doi: 10.1067/mod.2001.115616. PMID 11455373
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration. Center for Drug Evaluation and Research (CDER); Center for Biologics Evaluation and Research (CBER). Population Pharmacokinetics, Guidance for Industry. (February 2022). https://www.fda.gov/regulatory-information/search-fda-guidance-documents/population-pharmacokinetics
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration. Center for Drug Evaluation and Research (CDER). General Clinical Pharmacology Considerations for Pediatric Studies of Drugs, Including Biological Products. Guidance for Industry (Draft). (September 2022). https://www.fda.gov/regulatory-information/search-fda-guidance-documents/general-clinical-pharmacologyconsiderations- pediatric-studies-drugs-including-biological-products
- [Background] Wang Y, Jadhav PR, Lala M, Gobburu JV. Clarification on precision criteria to derive sample size when designing pediatric pharmacokinetic studies. J Clin Pharmacol. 2012 Oct;52(10):1601-6. doi: 10.1177/0091270011422812. Epub 2011 Dec 12. No abstract available. PMID 22162537